CLINICAL TRIAL: NCT05677776
Title: The Relationship Between Covid-19 and Pneumothorax in Patients Hospitalized With Covid-19 During the Pandemic
Status: Completed | Type: Observational
Sponsor: Erol Olcok Corum Training and Research Hospital (Other)
Responsible Party: Principal Investigator, HULYA TOPCU, MD, Principal Investigator, Erol Olcok Corum Training and Research Hospital
Other Study IDs: 2021-98
Record Dates: First submitted 2023-01-07; First posted 2023-01-10 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: COVID-19; Pneumothorax
Keywords: COVID-19; pneumothorax
MeSH Terms: conditions — COVID-19; Pneumothorax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is aimed to examine the retrospective features of covid-19 patients followed in our hospital with pneumothorax.

DETAILED DESCRIPTION:
It is aimed to examine the retrospective features of covid-19 patients followed in our hospital with pneumothorax. The files of covid-19 patients with pneumothorax were reviewed retrospectively. The radiological records and treatment protocols of the patients were reviewed. The results were evaluated in terms of its relationship with pneumothorax.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years
* covid-19 patient
* having a diagnosis of pneumothorax
* PCR test positive and lung tomography pneumonic involvement

Exclusion Criteria:

* PCR test negative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: over 18 years , PCR testin positive COVID-19 patients
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
relationship between covid-19 and pneumothorax | 1 year
  Inflammatory markers, C-reactive protein (CRP), lactate dehydrogenase (LDH), ferritin, D-dimer, procalcitonin, blood gas lactate, creatine kinase, white blood cells, baseline laboratory test results including WBC, lymphocyte, neutrophil counts, platelets, urea, creatinine, and neutrophil/lymphocyte ratio were documented for each patient.
  Respiratory support status, the fraction of inspired oxygen (FiO2), positive end-expiratory pressure (PEEP) values, tidal volume, and duration of the mechanical ventilator (MV) stay were determined.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal BOYACI, Study Chair — ÇorumTRH
Locations (1):
- Hulya TOPCU, Çorum, Turkey (Türkiye)